CLINICAL TRIAL: NCT01705639
Title: Does Melatonin Treatment Affect Glucose Tolerance Among Individuals With a Variant (rs10830963) of the Melatonin Receptor 1B (MTNR1B) Gene?
Brief Title: Melatonin and Glucose Tolerance Among Individuals With a Variant of the MTNR1B Gene
Acronym: MELAG
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Helsinki (Other)
Collaborators: Lund University (Other); Folkhalsan Research Center (Unknown)
Responsible Party: Principal Investigator, Tom Forsén, MD PhD, University of Helsinki
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: EudraCT-2011-005360-22
Record Dates: First submitted 2012-10-10; First posted 2012-10-12 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Glucose Tolerance
Keywords: diabetes; melatonin; glucose tolerance; sleep
MeSH Terms: conditions — Diabetes Mellitus | interventions — Melatonin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Melatonin (Experimental): melatonin 4mg od for 3 months
  Interventions: Drug: Melatonin

INTERVENTIONS:
Drug: Melatonin — All subjects receive the same dose of melatonin
  Other Names: Circadin

SUMMARY:
The effect of 3 months of melatonin 4mg treatment on glucose tolerance in different variants of the melatonin receptor 1B gene will be evaluated. The following will be done at 0 and 3 months:

* OGTT
* questionnaires about sleep and activity
* Actigraph
* Anthropometry
* Blood pressure

DETAILED DESCRIPTION:
http://www.sciencedirect.com/science/article/pii/S1550413116301607

ELIGIBILITY:
Inclusion Criteria:

* signed informed concent
* Known genotype for MTNR1B from the Botnia-ppp study
* Age 18-75 years

Exclusion Criteria:

* Diabetes
* Positive GAD-ab
* Sever dysregulated hypertension
* glaucoma
* severe coronary heart disease or arrythmias
* previous or ongoing severe ventricle or duodenal ulcer
* psychosis or anxiety disorder
* regular use of sleep pills, antidepressants or neuroleptics
* creatinine > 130 µmol/L
* elevated liver enzymes (ASAT, ALAT, ALP, GT, bilirubin) > 3 times reference value
* inability to sign informed concent
* other factor with according to the physician may affect treatment or results.
* participation in other clinical study
* allergy to melatonin or other substance in the capsule
* hereditary galactose intolerance or glucose/galactose malabsorption
* intention to become pregnant

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2012-11; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Glucose tolerance | 3 months
  Glucose tolerance is measured in OGTT: 0,30,60,90 and 120 minute values of glucose and insulin.

SECONDARY OUTCOMES:
sleep | 3 months
  monitoring of sleep with questionnaires and activity monitoring
Activity | 3 months
  Activity and sleep of the subjects is recorded with Actigraph at 0 and 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Leif Groop, Prof., Study Chair — University of Lund, University of Helsinki; Tiinamaija Tuomi, Docent, Study Director — Helsinki University Central Hospital; Bo Isomaa, Docent, Principal Investigator — Folkhalsan
Locations (2):
- Finland (2):
  - Botniacentret Jakobstad, Jakobstad
  - Vasa health care centre, Vaasa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tuomi T, Nagorny CLF, Singh P, Bennet H, Yu Q, Alenkvist I, Isomaa B, Ostman B, Soderstrom J, Pesonen AK, Martikainen S, Raikkonen K, Forsen T, Hakaste L, Almgren P, Storm P, Asplund O, Shcherbina L, Fex M, Fadista J, Tengholm A, Wierup N, Groop L, Mulder H. Increased Melatonin Signaling Is a Risk Factor for Type 2 Diabetes. Cell Metab. 2016 Jun 14;23(6):1067-1077. doi: 10.1016/j.cmet.2016.04.009. Epub 2016 May 12. PMID 27185156